CLINICAL TRIAL: NCT00990587
Title: Phase 1 Study Evaluating the Tolerance and Biologic Activity of Oral Ciclopirox Olamine in Patients With Relapsed or Refractory Hematologic Malignancy
Brief Title: Study Evaluating the Tolerance and Biologic Activity of Oral Ciclopirox Olamine in Patients With Relapsed or Refractory Hematologic Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPX V001
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-06

CONDITIONS: Hematologic Malignancy; Acute Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Myelodysplasia; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia; Hodgkin's Disease
Keywords: relapsed and refractory hematologic malignancy; ALL (acute lymphoid leukemia); CLL (chronic lymphoid leukemia); High risk myelodysplasia (MDS) with an IPSS (International Prognostic Scoring System) score >2.5; CML (chronic myelogenous leukemia) blast crisis; Relapsed or refractory acute myeloid leukemia (AML)
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hodgkin Disease; Recurrence; Leukemia, B-Cell; Blast Crisis | interventions — Ciclopirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ciclopirox Olamine (Experimental): Patients will take Ciclopirox Olamine at escalating doses depending on when they enter into the trial.
  Interventions: Drug: Ciclopirox Olamine

INTERVENTIONS:
Drug: Ciclopirox Olamine — Patients will take Ciclopirox Olamine at various doses depending on which dose level they come into the study at. Ciclopirox olamine will be administered orally as an aqueous suspension without food. The starting dose will be 5 mg/m2/day administered as a single dose daily for 5 days (one cycle). Once a MTD has been determined, the new patients that enter into the trial will then take it at that level.

SUMMARY:
This is an open-label, single arm study. Approximately 3-30 patients will be enrolled. Patients will receive Oral ciclopirox olamine (aqueous suspension), initial starting dose of 5 mg/m2/day administered as a single dose daily for 5 days. Three patients will initially be treated at each dose level in sequential cohorts. Dose escalation will continue for each subsequent cohort based on toxicity and plasma drug concentrations observed during the previous cohort. Dose escalation will continue until establishment of the maximum tolerated dose (MTD) has been met.

Patients who have demonstrated response to treatment, up to 6 total cycles of treatment may be administered. If additional cycles are warranted, ciclopirox olamine will be given at the same dose and frequency as the patient initially received.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Relapsed or refractory hematologic malignancies including AML, ALL, CLL, high risk myelodysplasia (International Prognostic Score >2.5), CML blast crisis, multiple myeloma, non-Hodgkin's lymphoma, and Hodgkin's lymphoma for which all potentially curative therapy options have been exhausted.
3. ECOG (Eastern Cooperative Oncology Group) performance status < 2.
4. Biochemical values within the following range:

   1. Serum creatinine < 2x upper limit of normal.
   2. Total bilirubin < 2x upper limit of normal, AST (asparatate aminotransferase) and ALT (alanine aminotransferase) < 5x upper limit of normal.
5. Ability to maintain adequate oral intake of medication.
6. Ability to understand and sign informed consent.
7. Toxicity from prior chemotherapy has resolved

Exclusion Criteria:

1. Uncontrolled systemic infection.
2. Uncontrolled intercurrent illness
3. Pregnant or breast feeding
4. Active CNS (central nervous system) disease
5. Neurologic symptoms related to intracurrent illnesses or unexplained causes
6. Psychiatric illness that would limit compliance with study
7. Receiving other systemic chemotherapy, other than hydroxyurea to control circulating blast counts, within 10 days of study entry. Hydroxyurea is permitted, however the dose must be stable and unchanged in the 7 days prior to initiation with ciclopirox olamine
8. Concurrent therapy with topical ciclopirox olamine.
9. Use of other investigational anti-cancer therapy within two weeks of study entry.
10. Use of oral or intravenous metal supplements including iron, copper, zinc and nickel.
11. Resting ejection fraction < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose-limiting toxicity, maximum tolerated dose, and recommended phase II dose of ciclopirox olamine. | 2 years
To evaluate maximum tolerated dose. | 2 years
To evaluate recommended phase II dose of ciclopirox olamine. | 2 years

SECONDARY OUTCOMES:
To determine the pharmacodynamic effects of ciclopirox olamine on survivin expression, and relate to the steady-state plasma concentrations of ciclopirox olamine. | 2 years
To determine the response rate of ciclopirox olamine. | 2 years
To characterize the pharmacokinetics (PK) of ciclopirox olamine in patients with relapsed or refractory hematologic malignancy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Minden, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Song S, Christova T, Perusini S, Alizadeh S, Bao RY, Miller BW, Hurren R, Jitkova Y, Gronda M, Isaac M, Joseph B, Subramaniam R, Aman A, Chau A, Hogge DE, Weir SJ, Kasper J, Schimmer AD, Al-awar R, Wrana JL, Attisano L. Wnt inhibitor screen reveals iron dependence of beta-catenin signaling in cancers. Cancer Res. 2011 Dec 15;71(24):7628-39. doi: 10.1158/0008-5472.CAN-11-2745. Epub 2011 Oct 18. PMID 22009536